CLINICAL TRIAL: NCT04936529
Title: Phase II Trial of a Bivalent Vaccine With the Immunological Adjuvant OPT-821 (QS-21), in Combination With Oral β-glucan and Randomization of GM-CSF, for High-risk Neuroblastoma
Brief Title: A Study of a Vaccine in Combination With β-glucan and GM-CSF in People With Neuroblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 21-206
Record Dates: First submitted 2021-06-16; First posted 2021-06-23 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; High-risk Neuroblastoma; OPT-821; QS-21; β-glucan; GM-CSF; Memorial Sloan Kettering Cancer Center; 21-206
MeSH Terms: conditions — Neuroblastoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; saponin QA-21V1

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Group 1 participants receive oral β-glucan (40 mg/kg/day x 14 days) starting week 1. This schedule includes annual booster vaccinations, with β-glucan, administered at weeks 8, 20, 32, 52, 78, 104, and 156 (vaccinations #1 & #4-10). Participants will not receive GM-CSF.
  Interventions: Dietary Supplement: β-glucan; Biological: OPT-821
- Group 2 (Experimental): Group 2 participants receive oral β-glucan (40 mg/kg/day) starting week 1. Participants also receive GM-CSF (250 mcg/m2/day) x3 days with vaccinations #1-#3; x7 days with vaccinations #4-#9; and x5 days with vaccination #10. The treatment includes annual booster vaccinations, with a 2-week cycle of β-glucan, administered at weeks 8, 20, 32, 52, 78, 104, and 156 (vaccinations #1 & #4-10)
  Interventions: Dietary Supplement: β-glucan; Drug: GM-CSF; Biological: OPT-821
- Group 3 (Experimental): Group 3 will include participants who cannot be randomized (e.g., due to allergy to GMCSF). It will also include participants previously treated with this vaccine and oral β-glucan on the predecessor MSK protocol IRB# 05-075 or on this protocol (participants can therefore be enrolled more than one time on this protocol). These participants will be treated as in Group 1. Participants who are registered to Group 3 and have been previously treated with vaccine (in this protocol or MSK predecessor 05-075) will not receive vaccines 4 and 6. These patients will receive a total of 8 injections. The analyses in this group will be exploratory.
  Interventions: Dietary Supplement: β-glucan; Biological: OPT-821

INTERVENTIONS:
Dietary Supplement: β-glucan — Group 1 participants receive oral β-glucan (40 mg/kg/day) starting week 1 and continue with ~2 weeks on, ~2 weeks off, up to 1 cycle after vaccination #7, then 1 cycle with each subsequent vaccination (#8-#14). This schedule includes annual booster vaccinations, with a 2-week cycle of β-glucan, administered at months 36 (3 years), 48 (4 years), and 60 (5 years).
  Group 2 participants receive oral β-glucan (40 mg/kg/day) starting week 1 and continue with ~2 weeks on, ~2 weeks off, up to 1 cycle after vaccination #7, then 1 cycle with each subsequent vaccination (#8-#14).
  Group 3 participants will be treated as in Group 1.
  Other Names: oral β-glucan
Drug: GM-CSF — Group 1 participants will not receive GM-CSF.
  Group 2 participants will receive GM-CSF (250 mcg/m2/day) x3 days with vaccinations #1-#3; x7 days with vaccinations #4-#11; and x5 days with vaccinations #12-#14.
  Group 3 participants will be treated as in Group 1.
  Arms: Group 2
Biological: OPT-821 — Vaccine injections must occur a minimum of 6 days apart. After the first four vaccine injections, vaccines can be administered up to two weeks earlier or later than indicated without representing a protocol violation.
  Other Names: QS-21

SUMMARY:
The purpose of the study is to explore the combination of a bivalent vaccine, a sugar called beta-glucan (β-glucan), and a protein called granulocyte-macrophage colony stimulating factor (GM-CSF) as an effective treatment for people with high-risk neuroblastoma that is in complete remission. The combination may be effective because the different parts of the treatment work to strengthen the immune system's response against cancer cells in different ways.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NB as defined by international criteria, i.e., histopathology (confirmed by the MSK Department of Pathology) or BM metastases plus high urine catecholamine levels or positivity in MIBG scan
* HR-NB as defined by risk-related treatment guidelines and international criteria,i.e., metastatic/non-localized disease with MYCN amplification (any age), MYCN-non-amplified metastatic disease >18 months old, MYCNamplified localized disease (any age), or disease resistant to standard chemotherapy.
* HR-NB (as defined above) and in 1) first CR at ≥ 6 months from initiation of immunotherapy using anti-GD2 antibody, or 2) second or subsequent CR (achieved after treatment for PD). CR is defined according to the International Neuroblastoma Response Criteria.Patients with positive MIBG scan but negative FDG-PET scan, and CR in BM, are eligible.
* Patients with grade 3 toxicities or less using the Common Toxicity Criteria (Version 5.0) developed by the National Cancer Institute of the USA (CTCAE v5.0) related to hematologic, cardiac, neurological, pulmonary, renal, hepatic or gastrointestinal function as determined by blood tests or physical exam.
* Hematologic Function

  * Absolute neutrophil count (ANC) ≥ 500/mcl
  * Absolute lymphocyte count ≥ 500/mcl
  * Hemaglobin (Hgb) ≥ 8 g/dL
  * Platelet count ≥ 50,000 mm^3
* Renal Function o Serum creatinine ≤ 3.0 x ULN

or

* eGFR >60 mL/min/1.73 m^2

  - Hepatic Function
* Serum bilirubin ≤ 3.0 × ULN
* Aspartate transaminase (AST) ≤ 5.0 × ULN
* Alanine aminotransferase (ALT) ≤ 5.0 × ULN

  * Prior treatment with other immunotherapy, including mAbs or vaccine, is allowed but must be completed ≥ 21 days before the 1st vaccination.

Note: Prior treatment with an investigational therapy must be completed ≥ 28 days before the 1st vaccination.

* ≥ 21 and ≤ 180 days between completion of systemic therapy and 1st vaccination.
* Patients have recovered from any toxicities grade 3 or higher caused by prior therapies.
* Patients previously enrolled on this trial are eligible for repeat enrollment if they did not complete all vaccine injections during the first time on protocol but they will be assigned to Group 3 and will not be included in the primary biostatistical analyses.
* A negative pregnancy test is required for patients w ith child-bearing capability.
* Signed informed consent indicating awareness of the investigational nature of this program.

Exclusion Criteria:

* Patients w ith significant (grade >4) hematologic, cardiac, neurological, pulmonary, renal, hepatic or gastrointestinal function as determined by blood tests or physical exam, using the Common Toxicity Criteria (Version 5.0) developed by the National Cancer Institute of the USA (CTCAE v5.0)
* History of allergy to KLH, QS-21, OPT-821, or glucan.
* Active life-threatening infection requiring systemic therapy.
* Inability to comply with protocol requirements.
* Patients with history of allergy to GM-CSF or who are unable to obtain GM-CSF because of insurance issues are ineligible

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2021-08-02 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Effect of GM-CSF on anti-GD2 antibody titers | 32 weeks
  Effect of GM-CSF on anti-GD2 antibody titers among patients who are in first or second (or later) CR, i.e., have no evidence of NB by standard studies.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kushner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org